CLINICAL TRIAL: NCT00518167
Title: The Finnish Diabetes Prevention Study: A Follow-up Study on the Effect of a Dietary and Exercise Intervention in the Prevention of Diabetes and Its Vascular Complications
Brief Title: The Finnish Diabetes Prevention Study
Acronym: DPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of Eastern Finland (Other); Finnish Diabetes Association (Other); University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KTL151-6
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; primary prevention; diet; physical activity; intervention; impaired glucose tolerance; lifestyle; randomized controlled study
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intensive lifestyle intervention
  Interventions: Behavioral: Intensive lifestyle counselling
- 2 (No Intervention): Standard counselling at baseline

INTERVENTIONS:
Behavioral: Intensive lifestyle counselling — Individualized dietary and physical activity counselling aiming at
  1. weight reduction
  2. dietary fibre 15 g /1000 kcal or more
  3. energy proportion of dietary fat less than 30%
  4. energy proportion of saturated fat less than 10%
  5. moderate physical activity >30 minutes per day or 4 hours per week
  Arms: 1

SUMMARY:
The aim of this study is to clarify whether lifestyle intervention provided to people with high type 2 diabetes risk will lower the cumulative incidence of diabetes. Furthermore, the aim is to study the effect of lifestyle intervention on cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance (p-glucose 2 hours after a 75 g oral glucose load between 7.8 and 11.0 mmol/l)
* body mass index 25 or higher

Exclusion Criteria:

* diabetes (previous gestational diabetes accepted)
* other chronic disease rendering survival for 6 years
* condition or medication affecting glucose tolerance
* recent myocardial infarction

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 1993-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diabetes incidence | During the intervention period + after the intervention has been stopped

SECONDARY OUTCOMES:
CVD incidence | During the total follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko Tuomilehto, professor emeritus, Principal Investigator — Finnish Institute for Health and Welfare and University of Helsinki; Matti Uusitupa, professor emeritus, Principal Investigator — University of Eastern Finland
Locations (4):
- Finland (4):
  - Population Health Unit, Department of Public Health and Welfare, Finnish Institute for Health and Welfare, Helsinki
  - Institute of Public Health and Clinical Nutrition, University of Eastern Finland, Kuopio
  - Department of Sports Medicine, Oulu Deaconess Institute, Oulu
  - The Diabetes Center, Finnish Diabetes Association, Tampere

REFERENCES:
- [Background] Eriksson J, Lindstrom J, Valle T, Aunola S, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Lauhkonen M, Lehto P, Lehtonen A, Louheranta A, Mannelin M, Martikkala V, Rastas M, Sundvall J, Turpeinen A, Viljanen T, Uusitupa M, Tuomilehto J. Prevention of Type II diabetes in subjects with impaired glucose tolerance: the Diabetes Prevention Study (DPS) in Finland. Study design and 1-year interim report on the feasibility of the lifestyle intervention programme. Diabetologia. 1999 Jul;42(7):793-801. doi: 10.1007/s001250051229. PMID 10440120
- [Background] Lindgren P, Lindstrom J, Tuomilehto J, Uusitupa M, Peltonen M, Jonsson B, de Faire U, Hellenius ML; DPS Study Group. Lifestyle intervention to prevent diabetes in men and women with impaired glucose tolerance is cost-effective. Int J Technol Assess Health Care. 2007 Spring;23(2):177-83. doi: 10.1017/S0266462307070286. PMID 17493303
- [Background] Laitinen T, Lindstrom J, Eriksson J, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M. Cardiovascular autonomic dysfunction is associated with central obesity in persons with impaired glucose tolerance. Diabet Med. 2011 Jun;28(6):699-704. doi: 10.1111/j.1464-5491.2011.03278.x. PMID 21388444
- [Result] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Result] Eriksson J, Valle T, Lindstrom J, Haffner S, Louheranta A, Uusitupa M, Tuomilehto J. Leptin concentrations and their relation to body fat distribution and weight loss--a prospective study in individuals with impaired glucose tolerance. DPS-study group. Horm Metab Res. 1999 Nov;31(11):616-9. doi: 10.1055/s-2007-978807. PMID 10598830
- [Result] Uusitupa M, Louheranta A, Lindstrom J, Valle T, Sundvall J, Eriksson J, Tuomilehto J. The Finnish Diabetes Prevention Study. Br J Nutr. 2000 Mar;83 Suppl 1:S137-42. doi: 10.1017/s0007114500001070. PMID 10889804
- [Result] Lindi VI, Uusitupa MI, Lindstrom J, Louheranta A, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Tuomilehto J; Finnish Diabetes Prevention Study. Association of the Pro12Ala polymorphism in the PPAR-gamma2 gene with 3-year incidence of type 2 diabetes and body weight change in the Finnish Diabetes Prevention Study. Diabetes. 2002 Aug;51(8):2581-6. doi: 10.2337/diabetes.51.8.2581. PMID 12145174
- [Result] Kubaszek A, Pihlajamaki J, Komarovski V, Lindi V, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study. Promoter polymorphisms of the TNF-alpha (G-308A) and IL-6 (C-174G) genes predict the conversion from impaired glucose tolerance to type 2 diabetes: the Finnish Diabetes Prevention Study. Diabetes. 2003 Jul;52(7):1872-6. doi: 10.2337/diabetes.52.7.1872. PMID 12829659
- [Result] Uusitupa M, Lindi V, Louheranta A, Salopuro T, Lindstrom J, Tuomilehto J; Finnish Diabetes Prevention Study Group. Long-term improvement in insulin sensitivity by changing lifestyles of people with impaired glucose tolerance: 4-year results from the Finnish Diabetes Prevention Study. Diabetes. 2003 Oct;52(10):2532-8. doi: 10.2337/diabetes.52.10.2532. PMID 14514637
- [Result] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Result] Todorova B, Kubaszek A, Pihlajamaki J, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study. The G-250A promoter polymorphism of the hepatic lipase gene predicts the conversion from impaired glucose tolerance to type 2 diabetes mellitus: the Finnish Diabetes Prevention Study. J Clin Endocrinol Metab. 2004 May;89(5):2019-23. doi: 10.1210/jc.2003-031325. PMID 15126514
- [Result] Laukkanen O, Pihlajamaki J, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study Group. Common polymorphisms in the genes regulating the early insulin signalling pathway: effects on weight change and the conversion from impaired glucose tolerance to Type 2 diabetes. The Finnish Diabetes Prevention Study. Diabetologia. 2004 May;47(5):871-7. doi: 10.1007/s00125-004-1395-6. Epub 2004 May 1. PMID 15127203
- [Result] Siitonen N, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M, Uusitupa M. Association between a deletion/insertion polymorphism in the alpha2B-adrenergic receptor gene and insulin secretion and Type 2 diabetes. The Finnish Diabetes Prevention Study. Diabetologia. 2004 Aug;47(8):1416-24. doi: 10.1007/s00125-004-1462-z. Epub 2004 Jul 28. PMID 15309292
- [Result] Ilanne-Parikka P, Eriksson JG, Lindstrom J, Hamalainen H, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Rastas M, Salminen V, Aunola S, Sundvall J, Valle T, Lahtela J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Prevalence of the metabolic syndrome and its components: findings from a Finnish general population sample and the Diabetes Prevention Study cohort. Diabetes Care. 2004 Sep;27(9):2135-40. doi: 10.2337/diacare.27.9.2135. PMID 15333474
- [Result] Salopuro T, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M, Uusitupa M. Common variants in beta2- and beta3-adrenergic receptor genes and uncoupling protein 1 as predictors of the risk for type 2 diabetes and body weight changes. The Finnish Diabetes Prevention Study. Clin Genet. 2004 Oct;66(4):365-7. doi: 10.1111/j.1399-0004.2004.00313.x. No abstract available. PMID 15355441
- [Result] Laukkanen O, Pihlajamaki J, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study Group. Polymorphisms of the SUR1 (ABCC8) and Kir6.2 (KCNJ11) genes predict the conversion from impaired glucose tolerance to type 2 diabetes. The Finnish Diabetes Prevention Study. J Clin Endocrinol Metab. 2004 Dec;89(12):6286-90. doi: 10.1210/jc.2004-1204. PMID 15579791
- [Result] Laaksonen DE, Lindstrom J, Lakka TA, Eriksson JG, Niskanen L, Wikstrom K, Aunola S, Keinanen-Kiukaanniemi S, Laakso M, Valle TT, Ilanne-Parikka P, Louheranta A, Hamalainen H, Rastas M, Salminen V, Cepaitis Z, Hakumaki M, Kaikkonen H, Harkonen P, Sundvall J, Tuomilehto J, Uusitupa M; Finnish diabetes prevention study. Physical activity in the prevention of type 2 diabetes: the Finnish diabetes prevention study. Diabetes. 2005 Jan;54(1):158-65. doi: 10.2337/diabetes.54.1.158. PMID 15616024
- [Result] Lindstrom J, Peltonen M, Tuomilehto J. Lifestyle strategies for weight control: experience from the Finnish Diabetes Prevention Study. Proc Nutr Soc. 2005 Feb;64(1):81-8. doi: 10.1079/pns2004412. PMID 15877926
- [Result] Laukkanen O, Lindstrom J, Eriksson J, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study. Polymorphisms in the SLC2A2 (GLUT2) gene are associated with the conversion from impaired glucose tolerance to type 2 diabetes: the Finnish Diabetes Prevention Study. Diabetes. 2005 Jul;54(7):2256-60. doi: 10.2337/diabetes.54.7.2256. PMID 15983230
- [Result] Salopuro T, Pulkkinen L, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M, Uusitupa M; Finnish Diabetes Prevention Study Group. Genetic variation in leptin receptor gene is associated with type 2 diabetes and body weight: The Finnish Diabetes Prevention Study. Int J Obes (Lond). 2005 Oct;29(10):1245-51. doi: 10.1038/sj.ijo.0803024. PMID 15997246
- [Result] Hamalainen H, Ronnemaa T, Virtanen A, Lindstrom J, Eriksson JG, Valle TT, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Rastas M, Aunola S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Improved fibrinolysis by an intensive lifestyle intervention in subjects with impaired glucose tolerance. The Finnish Diabetes Prevention Study. Diabetologia. 2005 Nov;48(11):2248-53. doi: 10.1007/s00125-005-1938-5. Epub 2005 Oct 5. PMID 16205886
- [Result] Niskanen L, Laaksonen DE, Lindstrom J, Eriksson JG, Keinanen-Kiukaanniemi S, Ilanne-Parikka P, Aunola S, Hamalainen H, Tuomilehto J, Uusitupa M. Serum uric acid as a harbinger of metabolic outcome in subjects with impaired glucose tolerance: the Finnish Diabetes Prevention Study. Diabetes Care. 2006 Mar;29(3):709-11. doi: 10.2337/diacare.29.03.06.dc05-1465. No abstract available. PMID 16505534
- [Result] Lindstrom J, Peltonen M, Eriksson JG, Louheranta A, Fogelholm M, Uusitupa M, Tuomilehto J. High-fibre, low-fat diet predicts long-term weight loss and decreased type 2 diabetes risk: the Finnish Diabetes Prevention Study. Diabetologia. 2006 May;49(5):912-20. doi: 10.1007/s00125-006-0198-3. Epub 2006 Mar 16. PMID 16541277
- [Result] Siitonen N, Pulkkinen L, Mager U, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M, Uusitupa M. Association of sequence variations in the gene encoding adiponectin receptor 1 (ADIPOR1) with body size and insulin levels. The Finnish Diabetes Prevention Study. Diabetologia. 2006 Aug;49(8):1795-805. doi: 10.1007/s00125-006-0291-7. Epub 2006 May 25. PMID 16724230
- [Result] Mager U, Lindi V, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M, Pulkkinen L, Uusitupa M; Finnish Diabetes Prevention Study Group. Association of the Leu72Met polymorphism of the ghrelin gene with the risk of Type 2 diabetes in subjects with impaired glucose tolerance in the Finnish Diabetes Prevention Study. Diabet Med. 2006 Jun;23(6):685-9. doi: 10.1111/j.1464-5491.2006.01870.x. PMID 16759313
- [Result] Herder C, Peltonen M, Koenig W, Kraft I, Muller-Scholze S, Martin S, Lakka T, Ilanne-Parikka P, Eriksson JG, Hamalainen H, Keinanen-Kiukaanniemi S, Valle TT, Uusitupa M, Lindstrom J, Kolb H, Tuomilehto J. Systemic immune mediators and lifestyle changes in the prevention of type 2 diabetes: results from the Finnish Diabetes Prevention Study. Diabetes. 2006 Aug;55(8):2340-6. doi: 10.2337/db05-1320. PMID 16873699
- [Result] Mager U, Kolehmainen M, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto JO, Pulkkinen L, Uusitupa MI; Finnish Diabetes Prevention Study Group. Association between ghrelin gene variations and blood pressure in subjects with impaired glucose tolerance. Am J Hypertens. 2006 Sep;19(9):920-6. doi: 10.1016/j.amjhyper.2006.02.017. PMID 16942934
- [Result] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Result] Laaksonen DE, Siitonen N, Lindstrom J, Eriksson JG, Reunanen P, Tuomilehto J, Uusitupa M; Finnish Diabetes Prevention Study Group. Physical activity, diet, and incident diabetes in relation to an ADRA2B polymorphism. Med Sci Sports Exerc. 2007 Feb;39(2):227-32. doi: 10.1249/01.mss.0000246998.02095.bf. PMID 17277585
- [Result] Ottelin AM, Lindstrom J, Peltonen M, Martikainen J, Uusitupa M, Gylling H, Poutanen K, Louheranta A, Mannelin M, Paturi M, Salminen V, Tuomilehto J; Finnish Diabetes Prevention Study Group. Costs of a self-selected, health-promoting diet among the participants of the Finnish Diabetes Prevention Study. Diabetes Care. 2007 May;30(5):1275-7. doi: 10.2337/dc06-2444. Epub 2007 Feb 26. No abstract available. PMID 17325262
- [Result] Wang J, Kuusisto J, Vanttinen M, Kuulasmaa T, Lindstrom J, Tuomilehto J, Uusitupa M, Laakso M. Variants of transcription factor 7-like 2 (TCF7L2) gene predict conversion to type 2 diabetes in the Finnish Diabetes Prevention Study and are associated with impaired glucose regulation and impaired insulin secretion. Diabetologia. 2007 Jun;50(6):1192-200. doi: 10.1007/s00125-007-0656-6. Epub 2007 Apr 17. PMID 17437080
- [Result] Tolppanen AM, Pulkkinen L, Kolehmainen M, Schwab U, Lindstrom J, Tuomilehto J, Uusitupa M; Finnish Diabetes Prevention Study Group. Tenomodulin is associated with obesity and diabetes risk: the Finnish diabetes prevention study. Obesity (Silver Spring). 2007 May;15(5):1082-8. doi: 10.1038/oby.2007.613. PMID 17495183
- [Result] Kilpelainen TO, Lakka TA, Laaksonen DE, Laukkanen O, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Aunola S, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M, Laakso M; Finnish Diabetes Prevention Study Group. Physical activity modifies the effect of SNPs in the SLC2A2 (GLUT2) and ABCC8 (SUR1) genes on the risk of developing type 2 diabetes. Physiol Genomics. 2007 Oct 22;31(2):264-72. doi: 10.1152/physiolgenomics.00036.2007. Epub 2007 Jul 17. PMID 17636114
- [Result] Uusitupa M, Peltonen M, Lindstrom J, Aunola S, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Valle TT, Eriksson JG, Tuomilehto J; Finnish Diabetes Prevention Study Group. Ten-year mortality and cardiovascular morbidity in the Finnish Diabetes Prevention Study--secondary analysis of the randomized trial. PLoS One. 2009 May 21;4(5):e5656. doi: 10.1371/journal.pone.0005656. PMID 19479072
- [Result] Pajunen P, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J, Lindstrom J; Finnish Diabetes Prevention Study. HbA(1c) in diagnosing and predicting Type 2 diabetes in impaired glucose tolerance: the Finnish Diabetes Prevention Study. Diabet Med. 2011 Jan;28(1):36-42. doi: 10.1111/j.1464-5491.2010.03183.x. PMID 21166843
- [Derived] Ibrahim MMA, Uusitupa M, Tuomilehto J, Lindstrom J, Kjellsson MC, Karlsson MO. Competing Risks Analysis of the Finnish Diabetes Prevention Study. CPT Pharmacometrics Syst Pharmacol. 2025 Sep;14(9):1459-1469. doi: 10.1002/psp4.70065. Epub 2025 Jun 30. PMID 40583490
- [Derived] Salmela J, Konttinen H, Lappalainen R, Muotka J, Antikainen A, Lindstrom J, Tuomilehto J, Uusitupa M, Karhunen L. Eating behavior dimensions and 9-year weight loss maintenance: a sub-study of the Finnish Diabetes prevention study. Int J Obes (Lond). 2023 Jul;47(7):564-573. doi: 10.1038/s41366-023-01300-w. Epub 2023 May 6. PMID 37149709
- [Derived] Kivela J, Meinila J, Uusitupa M, Tuomilehto J, Lindstrom J. Longitudinal Branched-Chain Amino Acids, Lifestyle Intervention, and Type 2 Diabetes in the Finnish Diabetes Prevention Study. J Clin Endocrinol Metab. 2022 Sep 28;107(10):2844-2853. doi: 10.1210/clinem/dgac463. PMID 35917829
- [Derived] Penn L, White M, Lindstrom J, den Boer AT, Blaak E, Eriksson JG, Feskens E, Ilanne-Parikka P, Keinanen-Kiukaanniemi SM, Walker M, Mathers JC, Uusitupa M, Tuomilehto J. Importance of weight loss maintenance and risk prediction in the prevention of type 2 diabetes: analysis of European Diabetes Prevention Study RCT. PLoS One. 2013;8(2):e57143. doi: 10.1371/journal.pone.0057143. Epub 2013 Feb 25. PMID 23451166
- [Derived] Lindstrom J, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS). Improved lifestyle and decreased diabetes risk over 13 years: long-term follow-up of the randomised Finnish Diabetes Prevention Study (DPS). Diabetologia. 2013 Feb;56(2):284-93. doi: 10.1007/s00125-012-2752-5. Epub 2012 Oct 24. PMID 23093136
- [Derived] de Mello VD, Lindstrom J, Eriksson J, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Sundvall J, Laakso M, Tuomilehto J, Uusitupa M. Insulin secretion and its determinants in the progression of impaired glucose tolerance to type 2 diabetes in impaired glucose-tolerant individuals: the Finnish Diabetes Prevention Study. Diabetes Care. 2012 Feb;35(2):211-7. doi: 10.2337/dc11-1272. Epub 2011 Dec 30. PMID 22210578
- [Derived] Siitonen N, Pulkkinen L, Lindstrom J, Kolehmainen M, Schwab U, Eriksson JG, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M. Association of ADIPOR2 gene variants with cardiovascular disease and type 2 diabetes risk in individuals with impaired glucose tolerance: the Finnish Diabetes Prevention Study. Cardiovasc Diabetol. 2011 Sep 24;10:83. doi: 10.1186/1475-2840-10-83. PMID 21943112
- [Derived] Siitonen N, Pulkkinen L, Lindstrom J, Kolehmainen M, Eriksson JG, Venojarvi M, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M. Association of ADIPOQ gene variants with body weight, type 2 diabetes and serum adiponectin concentrations: the Finnish Diabetes Prevention Study. BMC Med Genet. 2011 Jan 10;12:5. doi: 10.1186/1471-2350-12-5. PMID 21219602
- [Derived] Uusitupa MI, Stancakova A, Peltonen M, Eriksson JG, Lindstrom J, Aunola S, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Laakso M. Impact of positive family history and genetic risk variants on the incidence of diabetes: the Finnish Diabetes Prevention Study. Diabetes Care. 2011 Feb;34(2):418-23. doi: 10.2337/dc10-1013. Epub 2010 Oct 27. PMID 20980412
- [Derived] Ilanne-Parikka P, Laaksonen DE, Eriksson JG, Lakka TA, Lindstr J, Peltonen M, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Leisure-time physical activity and the metabolic syndrome in the Finnish diabetes prevention study. Diabetes Care. 2010 Jul;33(7):1610-7. doi: 10.2337/dc09-2155. Epub 2010 Apr 22. PMID 20413514
- [Derived] Tuomilehto H, Peltonen M, Partinen M, Lavigne G, Eriksson JG, Herder C, Aunola S, Keinanen-Kiukaanniemi S, Ilanne-Parikka P, Uusitupa M, Tuomilehto J, Lindstrom J; Finnish Diabetes Prevention Study Group. Sleep duration, lifestyle intervention, and incidence of type 2 diabetes in impaired glucose tolerance: The Finnish Diabetes Prevention Study. Diabetes Care. 2009 Nov;32(11):1965-71. doi: 10.2337/dc08-1980. Epub 2009 Aug 3. PMID 19651919
- [Derived] Herder C, Peltonen M, Koenig W, Sutfels K, Lindstrom J, Martin S, Ilanne-Parikka P, Eriksson JG, Aunola S, Keinanen-Kiukaanniemi S, Valle TT, Uusitupa M, Kolb H, Tuomilehto J; Finnish Diabetes Prevention Study Group. Anti-inflammatory effect of lifestyle changes in the Finnish Diabetes Prevention Study. Diabetologia. 2009 Mar;52(3):433-42. doi: 10.1007/s00125-008-1243-1. Epub 2009 Jan 8. PMID 19130041
- [Derived] Lindstrom J, Peltonen M, Eriksson JG, Aunola S, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS) Group. Determinants for the effectiveness of lifestyle intervention in the Finnish Diabetes Prevention Study. Diabetes Care. 2008 May;31(5):857-62. doi: 10.2337/dc07-2162. Epub 2008 Feb 5. PMID 18252900